CLINICAL TRIAL: NCT05909436
Title: A Phase I/II Study Evaluating the Safety, Tolerability and Preliminary Efficacy of GLS-012 Monotherapy and in Combination With GLS-010 in Patients With Advanced Solid Tumors After Progression on Standard Treatment (Triumph-01)
Brief Title: Immuno-Oncology Drugs GLS-012 Alone & in Combination GLS-010 Treating With Advanced Patients Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLS-012-11
Record Dates: First submitted 2023-05-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and expansion of GLS-012 monotherapy and combination with GLS-010 (Experimental)
  Interventions: Drug: GLS-012; Drug: GLS-010

INTERVENTIONS:
Drug: GLS-012 — In the dose escalation stage of GLS-012 monotherapy, RP2D will be determined. All subjects will receive GLS-012 intravenously Q3W.
  In the expansion stage of GLS-012 monotherapy, subjects will receive up to 17 doses of GLS-012 at the RP2D administered Q3W.
  In the dose escalation stage of GLS-012 combination with GLS-010, RP2D of GLS-012 in combination with a fixed-dose GLS-010 will be determined. All subjects will receive GLS-012 and GLS-010 intravenously Q3W.
  In the expansion stage of GLS-012 combination with GLS-010, subjects will receive up to 35 doses of GLS-012 at the RP2D and GLS-010 at a fixed dose administered Q3W.
Drug: GLS-010 — In the dose escalation stage of GLS-012 combination with GLS-010, RP2D of GLS-012 in combination with a fixed-dose GLS-010 will be determined. All subjects will receive GLS-012 and GLS-010 intravenously Q3W.
  In the expansion stage of GLS-012 combination with GLS-010, subjects will receive up to 35 doses of GLS-012 at the RP2D and GLS-010 at a fixed dose administered Q3W.

SUMMARY:
This is a phase I/II study to investigate the safety, tolerability, and preliminary efficacy of GLS-012 monotherapy and in combination with GLS-010 in subjects with advanced solid rumor after progression on standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to sign the informed consent form;
2. Aged 18-75 years, male or female;
3. Histologically confirmed diagnosis of a solid tumor;
4. Patients with advanced solid tumors after progression on standard treatment;
5. Subjects must have at least 1 measurable target lesion according to RECIST version 1.1；
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1；
7. Life expectancy more than 12 weeks;
8. Adequate organ function and bone marrow function as indicated by the screening assessments in the screening period;
9. Women of childbearing potential must use highly effective contraception during the study period and at least 6 months after the last study drug administration, and must have a negative blood pregnancy test within 3 days before study enrollment.

Exclusion Criteria:

1. Patients with irAEs of grade ≥ 3 in the previous immunotherapy, and the AEs of the last anti-tumor treatment have not recovered to grade ≤ 1, except for hypothyroidism/hyperthyroidism and dermatitis that have recovered to grade ≤ 2, and AEs with no safety risks judged by the investigators, for example, alopecia.
2. Patients with primary or secondary immunodeficiency, or patients who are receiving long-term systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before randomization.
3. Use of corticosteroids or other immunosuppressants for systemic treatment within 14 days before the first study drug administration;
4. Known central nervous system (CNS) metastases;
5. Patients with severe hypersensitivity to macromolecular protein preparations/monoclonal antibodies in the past.
6. Patients with other malignant tumors within 5 years before screening, except cured cervical carcinoma in situ and cured skin basal cell carcinoma.
7. Cardiac clinical symptoms or diseases that are not well controlled.
8. Known hereditary or acquired bleeding and thrombosis tendency.
9. Patients with congenital or acquired immunodeficiency disorders (such as HIV-infection), or a history of organ transplantation.
10. Patients complying with any of hepatitis B surface antigen (HBsAg) positive and HBV-DNA copies being more than 2500 copies/ml (or 500 IU/ml); or positive HCV-RNA;
11. Patients with poor compliance or other conditions that are not suitable to participate in the clinical trial, as considered by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose-Limiting Toxicity (DLT) and MTD in the dose escalation stage | Up to 21 days after the first dose
Number of participants with treatment-related adverse events of GLS-012 monotherapy and in combination with GLS-010 in the expansion stage as assessed by CTCAE V5.0 | Up to approximately 24 months

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of GLS-012 monotherapy and in combination with GLS-010 | Up to approximately 4.5 months
Elimination half-life (T1/2) of GLS-012 monotherapy and in combination with GLS-010 | Up to approximately 4.5 months
Objective response rate (ORR) | Up to approximately 24 months
Disease control rate (DCR) | Up to approximately 24 months
Preliminary anti-tumor activity: Duration of response (DOR), time to response (TTR), progression free survival (PFS), overall survival (OS) | Up to approximately 24 months
Duration of response (DOR) | Up to approximately 24 months
Time to response (TTR) | Up to approximately 24 months
Progression free survival (PFS) | Up to approximately 24 months
Overall survival (OS) | Up to approximately 24 months

OTHER OUTCOMES:
Receptor occupancy (RO) of GLS-012 in the dose escalation stage of GLS-012 monotherapy | Up to approximately 4.5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China